CLINICAL TRIAL: NCT00806767
Title: Phase II Study of Allogeneic Transplant of Hematopoietic Stem Cells From a Compatible Family Donor in the Treatment of Patients Over 55 Years With Hematological Malignancies
Brief Title: Fludarabine, Busulfan, and Antilymphocyte Globulin Followed by Donor Stem Cell Transplant in Treating Older Patients With Hematological Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000626779; IPC-2005-004; EUDRACT-2005-005051-17; IPC-T2A; INCA-RECF0452
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic | interventions — gamma-Globulins; Busulfan; fludarabine phosphate

INTERVENTIONS:
Biological: therapeutic immune globulin
Drug: busulfan
Drug: fludarabine phosphate
Procedure: allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy before a donor stem cell transplant using stem cells that closely match the patient's stem cells, helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving antilymphocyte globulin before transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well fludarabine, busulfan, and antilymphocyte globulin together with donor stem cell transplant works in treating older patients with hematological cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess non-relapse or progression-related mortality at 1 year in patients over 55 with hematological malignancies undergoing allogeneic hematopoietic stem cell transplantation from a matched related, filgrastim (G-CSF)-mobilized donor and treated with conditioning comprising fludarabine phosphate, busulfan, and anti-lymphocyte globulin.
* To assess the incidence of graft-versus-host disease in these patients.
* To assess the incidence of relapse in these patients.
* To assess cellular recovery in these patients.
* To assess myeloid and lymphocyte chimerism in these patients.

Secondary

* To study the usual clinical and biological aspects of the transplantation in these patients.
* To study the impact of the Charlson score and the suitability for allogeneic transplantation score on mortality and 1-year survival.
* To assess the quality of life (QLQ-C30) of these patients.
* To study the economic cost of transplantation from conditioning to 1 year post-transplant.
* To study the mobilization and collection of progenitor stem cells in the donors.
* To study the psychological impact of donating stem cells on the donors.

OUTLINE: This is a multicenter study.

* Conditioning: Patients receive fludarabine phosphate IV over 30 minutes on days -5 through -1, busulphan IV over 2 hours every 6 hours on days -4 and -3, and anti-lymphocyte globulin IV over 4 hours on days -2 and -1.
* Transplantation: Patients undergo allogeneic hematopoietic stem call transplantation on day 0.

Patients complete a quality of life survey (QLQ-C30). After completion of study treatment, patients are followed every month for 6 months and then every 3 months for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a hematological malignancy
* Candidate for an allogeneic hematopoietic stem cell transplantation
* Available HLA-identical related donor

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy > 6 months
* LVEF ≥ 40%
* DLCO ≥ 50%
* Creatinine clearance ≥ 30 mL/min
* Transaminases and/or bilirubin ≤ 2 times upper limit of normal (ULN)
* No other cancer within the past 5 years, except for basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No human T-cell leukemia virus type 1 positivity
* No HIV positivity
* No uncontrolled bacterial, viral, or fungal infection
* No contraindications to the study drugs
* No concurrent serious and uncontrolled disease

PRIOR CONCURRENT THERAPY:

* At least 1 month since prior participation in a clinical trial

Ages: 56 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Allogeneic hematopoietic stem cell transplant-related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Didier Blaise, MD — Institut Paoli-Calmettes
Locations (1):
- Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille, France